CLINICAL TRIAL: NCT05009186
Title: Changing of PSA With Covid-19
Brief Title: Changing of Prostate Specific Antigen Value in Patients With Covid-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Omer Gokhan Doluoglu, Ankara Training and Research Hospital, Saglik Bilimleri Universitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSA
Record Dates: First submitted 2021-08-15; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Prostate Specific Antigen
Keywords: Covid-19; Prostate cancer; Prostate Specific Antigen
MeSH Terms: conditions — COVID-19; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: We measured PSA value during and after Covid-19 infection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Covid-19 group (Other): We will measure the PSA value during and after Covid-19 infection in the same group via paired simple t test
  Interventions: Other: PSA value

INTERVENTIONS:
Other: PSA value — We measure PSA value during and after covid-19 infection

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) caused a worldwide pandemic in over 100 years. The disease caused by this newly discovered virus was called Covid-19. In this study, we aimed to evaluate changing of PSA value in patients with Covid-19.

DETAILED DESCRIPTION:
Patients with positive PCR test results were included in the study. The age of the patient and urea, leukocyte, hemoglobin, platelet, urea, and creatinine values of the patients were recorded. Urinalysis and urine culture were taken from all patients. Acute phase reactants such as sedimentation, C-reaktif protein (CRP), ferritin, and fibrinogen were measured both at the time the patients applied and three weeks after the patient recovered. PSA and free PSA were also measured in the same way. Patients whose symptoms improved and the PCR test result was negative were considered as recovered.

ELIGIBILITY:
Inclusion Criteria:

* Male patients (>45 and <70 years of age) positive PCR test results were included in the study

Exclusion Criteria:

* The patients <45 and >70 years of age who described lower urinary tract symptoms who had urinary tract infection who a history of prostate biopsy and previous high level of PSA who history of prostatitis were excluded.

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The male patients >45 and <70 years of age included to the study
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
PSA value | 2 months
  prostate specific antigen

SECONDARY OUTCOMES:
Ferritin, CRP | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Omer G Doluoglu, Associate Professor, Principal Investigator — Ankara Training and Research Hospital
Locations (1):
- Omer Gokhan Doluoglu, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided